CLINICAL TRIAL: NCT00009984
Title: Randomized Phase II Study of Thalidomide Versus Thalidomide Plus Fludarabine for Patients With Chronic Lymphocytic Leukemia Previously Treated With Fludarabine
Brief Title: Thalidomide With or Without Fludarabine in Treating Patients With Hematologic Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02393; NYWCCC-MTS-00-0535ME; CDR0000068429; NCI-639; N01CM62204 (NIH)
Record Dates: First submitted 2001-02-02; First posted 2003-01-27 (Estimated); Last update posted 2013-06-06 (Estimated); Status verified 2013-06

CONDITIONS: Recurrent Small Lymphocytic Lymphoma; Refractory Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — fludarabine phosphate; Thalidomide

ARMS (2):
- Arm I (thalidomide) (Experimental): Patients receive oral thalidomide once daily in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: thalidomide
- Arm II (thalidomide, fludarabine phosphate) (Experimental): Patients receive thalidomide as in arm I and fludarabine IV over 30 minutes on days 1-5. Treatment with fludarabine repeats every 28 days for 6 courses. Once fludarabine is completed, patients continue to receive thalidomide alone as in arm I.
  Interventions: Drug: fludarabine phosphate; Drug: thalidomide

INTERVENTIONS:
Drug: fludarabine phosphate — Given IV
  Other Names: 2-F-ara-AMP; Beneflur; Fludara
  Arms: Arm II (thalidomide, fludarabine phosphate)
Drug: thalidomide — Given orally
  Other Names: Kevadon; Synovir; THAL; Thalomid

SUMMARY:
This randomized phase II trial is studying thalidomide and fludarabine to see how well they work compared to thalidomide alone in treating patients with hematologic cancer that has not responded to previous treatment with fludarabine. Thalidomide may stop the growth of hematologic cancer by stopping blood flow to the cancer. Combining thalidomide with fludarabine may increase the effectiveness of chemotherapy by making cancer cells more sensitive to the drug. It is not yet known whether thalidomide is more effective with or without fludarabine for hematologic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Compare the safety and tolerability of thalidomide with or without fludarabine in patients with fludarabine-refractory chronic lymphocytic leukemia or small lymphocytic lymphoma.

II. Compare the incidence of complete and partial remission in patients treated with these regimens.

OUTLINE: This is a randomized, open-label study. Patients are stratified according to time to relapse from last fludarabine treatment (less than 6 months vs more than 6 months). Patients are randomized to one of two treatment arms.

Arm I: Patients receive oral thalidomide once daily in the absence of disease progression or unacceptable toxicity.

Arm II: Patients receive thalidomide as in arm I and fludarabine IV over 30 minutes on days 1-5. Treatment with fludarabine repeats every 28 days for 6 courses. Once fludarabine is completed, patients continue to receive thalidomide alone as in arm I.

PROJECTED ACCRUAL: A total of 24-70 patients (12-35 per treatment arm) will be accrued for this study within 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of one of the following:

  * Confirmed chronic lymphocytic leukemia (CLL), meeting the following criteria:

    * Peripheral blood lymphocytosis greater than 5,000/mm^3
    * Co-expression of the CD5, CD19, CD20, and CD23 surface antigens
    * Clonal kappa and lambda light chain expression
    * Dim surface immunoglobulin expression
  * Small lymphocytic lymphoma
* Relapsed or refractory disease

  * Must have received at least 1 prior regimen containing fludarabine
  * Meets one of the following criteria:

    * Recurrence of lymphocytosis greater than 5,000/mm^3 or an increase in lymph node volume greater than 50% after achieving complete (CR) or partial response (PR)
    * Never achieved a CR or PR after receiving at least 2 courses of fludarabine IV for 5 days at a dose of 25 mg/m^2/day
* No other lymphoproliferative diseases or diseases due to transformation of CLL (e.g., prolymphocytic leukemia or Richter's syndrome)
* No known CNS disease
* Performance status - Karnofsky 60-100%
* At least 12 weeks
* See Disease Characteristics
* Bilirubin < 2.0 times upper limit of normal (ULN)*
* SGOT < 2.5 times ULN*
* Creatinine < 1.5 times ULN
* No history of cardiac arrhythmia
* No myocardial infarction within the past 6 months
* No other malignancy within the past 5 years except basal cell skin cancer or carcinoma in situ of the cervix
* No active serious infection uncontrolled by antibiotics
* No pre-existing neurotoxicity grade 3 or greater
* No other medical condition that would preclude study participation
* Not pregnant or nursing
* Negative pregnancy test
* Female patients must use 2 effective methods (at least 1 highly active method) of contraception 4 weeks before, during, and for 4 weeks after study participation and male patients must use effective barrier contraception during and for 4 weeks after study participation
* At least 4 weeks since prior biologic therapy and recovered
* No concurrent growth factors (epoetin alfa, filgrastim [G-CSF], or sargramostim [GM-CSF])
* See Disease Characteristics
* No more than 3 prior chemotherapy regimens
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas) and recovered
* No other concurrent chemotherapy
* At least 4 weeks since prior radiotherapy and recovered
* No concurrent radiotherapy
* Recovered from any prior investigational agents
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2002-03; Primary Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Toxicities graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v3.0 | Up to 5 years
Incidence of complete and partial remission | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Richard Furman, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States